CLINICAL TRIAL: NCT06406140
Title: Potential Effect of Niacin on Lipoprotein (a) Concentration and Hyperphosphatemia in End-Stage Renal Disease Patients Undergoing Hemodialysis
Brief Title: Study the Effect of Niacin on Lipoprotein (a) Concentration and Hyperphosphatemia in Hemodialysis Patients
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Amira Reda Muhammad Galal, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Interventional clinical study
Record Dates: First submitted 2024-04-19; First posted 2024-05-09 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-07

CONDITIONS: End-stage Renal Disease
Keywords: Hemodialysis; Niacin; Lipoprotein a
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Niacin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups each group includes 25 patients:
  Control group: 25 patients will receive their standard therapy only. Intervention group (niacin group): 25 patients will receive niacin 500 mg per day with their standard therapy for 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Niacin group (Experimental): patients will receive niacin-tablets 500 mg per day with their standard therapy for 3 months.
  Interventions: Drug: Niacin tablets 500 mg
- control group (No Intervention): patients will receive their standard therapy only

INTERVENTIONS:
Drug: Niacin tablets 500 mg — tablets used to treat hyperphosphatemia and lower lipoprotein a concentration in End-Stage Renal Disease Patients Undergoing Hemodialysis
  Other Names: Niacin 500 mg
  Arms: Experimental Niacin group

SUMMARY:
The goal of this clinical trial is to learn if Niacin has an effect on lipoprotein (a) concentration and hyperphosphatemia, which represent strong risk factors for cardiovascular diseases, in End-stage renal disease (ESRD) patients undergoing hemodialysis. It will also learn about the safety of Niacin. The main questions it aims to answer are:

* Does Niacin lower lipoprotein (a) concentration?
* Does Niacin treat hyperphosphatemia in End-stage renal disease (ESRD) patients undergoing hemodialysis? Researchers will compare Niacin to a control group (taking no drug) to see if drug Niacin works to treat hyperphosphatemia and lower lipoprotein (a) concentration.

Participants will:

* Take drug Niacin or no drug every day for 3 months
* Visit the clinic once every 2 weeks for checkups and tests

All Patients will be subjected to the following:

1. Informed consent.
2. Demographics and history taking: Using Patient Data sheet.
3. Laboratory evaluation including:

Kidney function tests: blood urea,serum creatinine, albumin ,uric acid. Complete blood count (CBC). Lipid profile:Lipoprotein (a),total cholesterol,triglyceride,high density lipoprotein (HDL), low density lipoprotein (LDL).

Phosphorous, calcium, sodium, parathyroid hormone (PTH), alkaline phosphatase (ALP).

C-reactive protein (CRP).

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a clinical syndrome secondary to the definitive change in function and/or structure of the kidney and is characterized by its irreversibility and slow and progressive evolution. CKD is very prevalent in the general adult population .End-stage renal disease (ESRD) was defined as a need for renal replacement therapy, CKD stage G5 (estimated glomerular filtration rate ≤ 15 mL/min per 1.73 m2) .Niacin (generic name of nicotinic acid), also known as vitamin B3, is a naturally occurring water-soluble vitamin that is essential in different biological activities. The active phosphate transport inhibitors are the newest interesting agents in the management of hyperphosphatemia alone or as add-on therapy to the existing phosphate binders. Niacin is one of this novel drug classes that has been demonstrated to show promising therapeutic potential in the treatment of hyperphosphatemia in HD patients.The aim of this study is to evaluate the effect of administration of niacin on lipoprotein (a) concentration and hyperphosphatemia, which represent strong risk factors for cardiovascular diseases, in ESRD patients undergoing hemodialysis.Patients will be randomized into two groups each group includes 25 patients:

Control group: 25 patients will receive their standard therapy only. Intervention group (niacin group): 25 patients will receive niacin 500 mg per day with their standard therapy for 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with ESRD, on maintenance hemodialysis for at least three (3) months.
2. Aged 18 years or older.
3. Both sexes.
4. No known contraindications to therapy with niacin.
5. Patients who accept to participate in the study.

Exclusion Criteria:

1. Pregnant and breast-feeding women
2. Any patient with a medical condition or taking any medications that would be contraindicated with the use of extended release niacin, such as active peptic ulcer disease;
3. History of severe allergic reactions to the study medication.
4. History of active infection or acute gouty attack within 2 weeks prior to enrollment;
5. Current medication regimen including niacin.
6. Chronic liver disease
7. Patients who had received immunosuppressive therapy
8. Non-compliant patients: those who did not adhere to the medications during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in serum phosphorus level | 3 months
  Niacin is expected to lower serum phosphorus levels in dialysis patients

SECONDARY OUTCOMES:
change in Lipoprotein (a) Concentration | 3 months
  Lipoprotein (a) , which has been suggested to play a role as an independent risk factor for coronary heart disease, is expected to be decreased by niacin

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab AlKasaby, professor, Principal Investigator — Dean of Faculty of Pharmacy (Girls), Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galal ARM, Salah MAR, Binsaleh AY, Alsubaie N, Alrossies AS, Elthakaby AH, Elsawy GM, Ali AA, Zalat ZAK. Targeting cardiovascular and metabolic risk modification in end stage renal disease (ESRD): a randomized controlled clinical trial on niacin's effects on lipoprotein(a) and biochemical markers in hemodialysis patients. Front Med (Lausanne). 2025 Oct 9;12:1625417. doi: 10.3389/fmed.2025.1625417. eCollection 2025. PMID 41140700